CLINICAL TRIAL: NCT03636100
Title: Systemic Release of Acetylcholine From the Autonomic Ganglionated Plexus: a Proposed Mechanism of Induced Hypotension During the Thaw Phase of Cryoballon Pulmonary Vein Ablation (GP RESPONSE Study)
Brief Title: Release of Acetylcholine From the Ganglionated Plexus During the Thaw Phase of Cryoballon Pulmonary Vein Ablation (GP RESPONSE Study)
Status: Terminated | Type: Observational
Why Stopped: After enrollment of half the subjects, the trial was unlikely to yield results
Sponsor: Saint Luke's Health System (Other)
Responsible Party: Sponsor
Other Study IDs: GP Response
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Catheter ablation; Cryoballon ablation; Acetylcholine; Ganglionated plexus; Pulmonary veins; Pulmonary vein isolation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Cryoballoon ablation — Cryoballoon ablation using standard equipment and techniques

SUMMARY:
Determine whether the presence of acetylcholine in the systemic circulation, correlates with the hypotensive response observed during the thaw phase of cryoballoon ablation.

DETAILED DESCRIPTION:
This will be a two-phase (feasibility and primary study phases), prospective observational study with pulmonary vein ablation applications during which a hypotensive response is not observed serving as within-subject controls. A total of 14 patients age 18-80 with atrial fibrillation undergoing first time cryoballoon ablation will be enrolled. Exclusion criteria are any prior left atrial ablation or cardiac surgery, a hemoglobin level of < 12.0 g/dL, or refusal or inability to provide informed consent.

The ablation procedure will be carried out per routine clinical practice by one operator. Two cryoballoon applications targeting 180 seconds per application will be performed per vein. Applications may be abbreviated at the discretion of the operator for indications such as balloon temperatures reaching the mid -50s C, esophageal temperatures approaching 20 C, or a decrease in diaphragmatic movement during phrenic nerve pacing. Application times may be extended to 200 to 240 seconds, also at the discretion of the operator, if within-freeze target temperatures (such as -30 C by 30 seconds or -40 C by 60 seconds) are not met.

A hypotensive response will be defined as a transient ≥ 20% decrease in systolic blood pressure from baseline (start of thaw) during the thaw phase and up to 60 seconds post-end of thaw (balloon deflation). A partial hypotensive response will be defined as a transient 10-19% decrease in systolic blood pressure. For all patients, the time from the end of the cryoballoon freeze to the end of the thaw, to the onset of the hypotensive response, and to blood pressure recovery within 10% of baseline will be recorded. Blood pressure and heart rate will be recorded at each time point. For the first 4 patients (phase I), blood samples of 2-3mL each will be drawn from the mid-right atrium at baseline and then at 30, 60 and 90 seconds after the end of each cryoballoon freeze application. Samples will also be drawn at onset of hypotension and 30 seconds later (superseding the drawing of other samples in the first 90 seconds post-end of freeze), and at blood pressure recovery. Samples will be drawn within 10 seconds of each specified time point; or will not be obtained and will be marked as a missing data point. If more than 20% of the specified data are missing for a given subject, that subject will be excluded from analysis. The samples will then be run on a commercially available 96-well colorimetric assay kit by Cell Biolabs Inc (catalog number STA-603) to assay for acetylcholine.

If the first phase of the study demonstrates the presence of acetylcholine at one or more time points during the thaw phase of 20% or more of cryoballoon applications during which a hypotensive response is observed, the study will proceed to phase 2. The results will be used to determine the optimal time point(s) at which to obtain samples during the second phase of the study (remaining 10 patients), with an anticipated need for 2-4 samples per cryoballoon application, one at start of thaw, another at a determined time point, and when there is a hypotensive response at the onset of hypotension and at blood pressure recovery. An interim report will be produced detailing the observations of phase 1 and specifying the plan for obtaining samples in phase 2.

ELIGIBILITY:
Inclusion Criteria:

* patients with atrial fibrillation undergoing first time cryoballoon ablation
* age 18-80

Exclusion Criteria:

* any prior left atrial ablation or cardiac surgery
* hemoglobin level of <12.0 g/dL
* refusal or inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 14 patients age 18-80 with atrial fibrillation undergoing first time cryoballoon ablation will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
Individual acetylcholine levels | 1 day
  With each subject serving as their own control, acetylcholine levels between ablation applications will be compared followed by a hypotensive response vs those that are not using paired T-tests.

SECONDARY OUTCOMES:
Group acetylcholine levels | 1 day
  Acetylcholine levels will be compared for the entire study group for applications followed by a hypotensive response vs those that are not. For this analysis each application will be treated as an independent unit and independent T-test will be used to compare acetylcholine levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Luke's Mid America Heart Institute, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrade J, Khairy P, Dobrev D, Nattel S. The clinical profile and pathophysiology of atrial fibrillation: relationships among clinical features, epidemiology, and mechanisms. Circ Res. 2014 Apr 25;114(9):1453-68. doi: 10.1161/CIRCRESAHA.114.303211. PMID 24763464
- [Background] Kojodjojo P, O'Neill MD, Lim PB, Malcolm-Lawes L, Whinnett ZI, Salukhe TV, Linton NW, Lefroy D, Mason A, Wright I, Peters NS, Kanagaratnam P, Davies DW. Pulmonary venous isolation by antral ablation with a large cryoballoon for treatment of paroxysmal and persistent atrial fibrillation: medium-term outcomes and non-randomised comparison with pulmonary venous isolation by radiofrequency ablation. Heart. 2010 Sep;96(17):1379-84. doi: 10.1136/hrt.2009.192419. PMID 20801856
- [Background] Nakagawa H, Scherlag BJ, Patterson E, Ikeda A, Lockwood D, Jackman WM. Pathophysiologic basis of autonomic ganglionated plexus ablation in patients with atrial fibrillation. Heart Rhythm. 2009 Dec;6(12 Suppl):S26-34. doi: 10.1016/j.hrthm.2009.07.029. Epub 2009 Oct 24. PMID 19959140
- [Background] Ketels S, Houben R, Van Beeumen K, Tavernier R, Duytschaever M. Incidence, timing, and characteristics of acute changes in heart rate during ongoing circumferential pulmonary vein isolation. Europace. 2008 Dec;10(12):1406-14. doi: 10.1093/europace/eun287. Epub 2008 Oct 19. PMID 18936041
- [Background] Peyrol M, Barraud J, Koutbi L, Maille B, Trevisan L, Martinez E, Levy S, Paganelli F, Franceschi F. Vagal Reactions during Cryoballoon-Based Pulmonary Vein Isolation: A Clue for Autonomic Nervous System Modulation? Biomed Res Int. 2016;2016:7286074. doi: 10.1155/2016/7286074. Epub 2016 May 3. PMID 27243034
- [Background] Lemery R. Bradycardia with cooling and cryo: A reminder of the autonomic effects of cold stimuli on the heart. Heart Rhythm. 2016 May;13(5):1018-1019. doi: 10.1016/j.hrthm.2015.12.049. Epub 2016 Jan 6. No abstract available. PMID 26767424
- [Background] Bordignon S, Furnkranz A, Dugo D, Perrotta L, Gunawardene M, Bode F, Klemt A, Nowak B, Schulte-Hahn B, Schmidt B, Chun KR. Improved lesion formation using the novel 28 mm cryoballoon in atrial fibrillation ablation: analysis of biomarker release. Europace. 2014 Jul;16(7):987-93. doi: 10.1093/europace/eut400. Epub 2014 Jan 19. PMID 24446511
- [Background] Yanagisawa S, Inden Y, Mizutani Y, Fujii A, Kamikubo Y, Kanzaki Y, Ando M, Funabiki J, Murase Y, Takenaka M, Otake N, Hattori T, Shibata R, Murohara T. Vagal response in cryoballoon ablation of atrial fibrillation and autonomic nervous system: Utility of epicardial adipose tissue location. J Arrhythm. 2017 Aug;33(4):275-282. doi: 10.1016/j.joa.2017.03.001. Epub 2017 Apr 24. PMID 28765757
- [Background] Kellogg DL Jr, Zhao JL, Coey U, Green JV. Acetylcholine-induced vasodilation is mediated by nitric oxide and prostaglandins in human skin. J Appl Physiol (1985). 2005 Feb;98(2):629-32. doi: 10.1152/japplphysiol.00728.2004. PMID 15649880
- [Background] Sun L, Dong JZ, DU X, Bai R, Li S, Salim M, Ma CS. Prophylactic Atropine Administration Prevents Vasovagal Response Induced by Cryoballoon Ablation in Patients with Atrial Fibrillation. Pacing Clin Electrophysiol. 2017 May;40(5):551-558. doi: 10.1111/pace.13072. Epub 2017 Apr 25. PMID 28295425
- [Background] Kuck KH, Furnkranz A, Chun KR, Metzner A, Ouyang F, Schluter M, Elvan A, Lim HW, Kueffer FJ, Arentz T, Albenque JP, Tondo C, Kuhne M, Sticherling C, Brugada J; FIRE AND ICE Investigators. Cryoballoon or radiofrequency ablation for symptomatic paroxysmal atrial fibrillation: reintervention, rehospitalization, and quality-of-life outcomes in the FIRE AND ICE trial. Eur Heart J. 2016 Oct 7;37(38):2858-2865. doi: 10.1093/eurheartj/ehw285. Epub 2016 Jul 5. PMID 27381589
- [Background] Kuck KH, Brugada J, Furnkranz A, Metzner A, Ouyang F, Chun KR, Elvan A, Arentz T, Bestehorn K, Pocock SJ, Albenque JP, Tondo C; FIRE AND ICE Investigators. Cryoballoon or Radiofrequency Ablation for Paroxysmal Atrial Fibrillation. N Engl J Med. 2016 Jun 9;374(23):2235-45. doi: 10.1056/NEJMoa1602014. Epub 2016 Apr 4. PMID 27042964
- [Background] Kampaktsis PN, Oikonomou EK, Y Choi D, Cheung JW. Efficacy of ganglionated plexi ablation in addition to pulmonary vein isolation for paroxysmal versus persistent atrial fibrillation: a meta-analysis of randomized controlled clinical trials. J Interv Card Electrophysiol. 2017 Dec;50(3):253-260. doi: 10.1007/s10840-017-0285-z. Epub 2017 Sep 8. PMID 28887742